CLINICAL TRIAL: NCT00090493
Title: UARK 2003-26, A Pilot Study of MAGE-A3 and NY-ESO-1 Immunotherapy in Combination With DTPACE Chemotherapy and Autologous Transplantation in Multiple Myeloma
Brief Title: Study of MAGE-A3 and NY-ESO-1 Immunotherapy in Combo With DTPACE Chemo and Auto Transplantation in Multiple Myeloma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2003-26
Record Dates: First submitted 2004-08-26; First posted 2004-08-31 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Mage-A3; Transplant; Peptide; DTPACE; vaccines; Immunotherapy; NY-ESO-1
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — MAGEA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MAGE-A3 and NY-ESO-1 Immunotherapy (Experimental): Treatment will consist of receiving peptide vaccinations as a shot just under the skin (subcutaneous). Peptides are small pieces of proteins. We have chosen to vaccinate with peptides derived from cancer proteins found in myeloma and other cancers. The purpose is to generate anti-myeloma T-cells which will kill myeloma cells and nothing else.
  Interventions: Biological: MAGE-A3; Biological: MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY

INTERVENTIONS:
Biological: MAGE-A3 — vaccinations at 2- week intervals (days 22,36,50) with the MAGE-A3 or NY-ESO-1 peptide and GM-CSF adjuvant. The peptides will be given s.c. in a dose of 300μg; GM-CSF (250μg) will be administered to promote attraction, maturation and longevity of DCs. #2 will be thawed and re-infused after transplant on day 81 and any anti-myeloma T-cells in this leukapheresis product will be boosted immediately by re-vaccinating the patient 3 times at 14 day intervals (vaccination #4-6: days 82, 96, and 110). Vaccines #4-6 will be identical to vaccines 1-3. Thereafter, 6 monthly vaccines will be given to further boost the anti-MM-T-cells.
Biological: MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY — Three injections with 300µg per injection (in 1.5mls) of peptide will be given subcutaneously together with the adjuvant GM-CSF at 500µg (same site in 0.5 mls) at two-week intervals

SUMMARY:
The hope is that the peptide vaccines will stimulate the immune system to attack and kill the myeloma cells. The purpose is to generate anti-myeloma T-cells which will kill myeloma cells and nothing else.

DETAILED DESCRIPTION:
This is an experimental treatment that will consist of receiving peptide vaccinations as a shot just under the skin (subcutaneous). We have chosen to vaccinate with peptides derived from cancer proteins found in myeloma and other cancers. The purpose is to generate anti-myeloma T-cells which will kill myeloma cells and nothing else.

The peptides are fragments from two tumor proteins called MAGE-A3 and NY-ESO-1. In order to be eligible for the study your myeloma cells must express either MAGE-A3 or NY-ESO-1, and your myeloma must be severe enough to require chemotherapy and stem cell transplantation. You must also have the appropriate HLA tissue type.

Patients who have MAGE-A3 positive myeloma and are HLA-A*0101 or -B*35 positive will receive the MAGE-A3 peptide vaccine.

Patients who have NY-ESO-1 positive myeloma and are HLA-A*0201 will receive the NY-ESO-1 peptide vaccine.

Three injections with 300µg per injection (in 1.5mls) of peptide will be given subcutaneously together with the adjuvant GM-CSF at 500µg (same site in 0.5 mls) at two-week intervals.

Your myeloma cells, obtained from a routine bone marrow aspirate, will be tested in the laboratory for the presence of MAGE-A3 and/or NY-ESO-1 proteins. HLA tissue type will be determined by standard methods in our Clinical Laboratory. This allows allocation of the correct vaccine to each individual patient.

Prior to starting a 6-day course of chemotherapy called DTPACE, white blood cells will be collected by a procedure called leukapheresis (leukapheresis no.1). Your white blood cells will be frozen for the duration of the chemotherapy in order to protect these white blood cells from the harmful effects of chemotherapy. After the chemotherapy is given, stem cells will be collected by leukapheresis (PBSC collection) and stored until the time of transplantation. After a short period of rest, the white blood cells from leukapheresis no.1 will be thawed and re-infused. This will ensure that you will have white blood cells that are in the best possible condition to respond to the peptide vaccines. A set of three vaccinations with the peptides at two-week intervals will follow. The hope is that the vaccinations will have generated precious anti-myeloma white blood cells.

You will again undergo leukapheresis (leukapheresis no.2) to collect the anti-myeloma white blood cells, which will be frozen in order to protect these precious cells from the chemotherapy drugs that will be infused just before the single or double auto-transplant.

A single dose of Melphalan will precede each transplant. The stem cells that were collected after DTPACE will be given for the transplants. For those receiving two transplants, a regimen of thalidomide with dexamethasone will be given for approximately 10 weeks between the two transplants. You will stop your thalidomide 28 days before the second transplant.

After completion of the transplants, the anti-myeloma white blood cells collected with leukapheresis no. 2 will be thawed and re-infused. These anti-myeloma cells will be boosted by three further peptide vaccinations at two-week intervals.

Finally, after you have completed these three vaccinations you will undergo another leukapheresis (no. 3). The anti-myeloma white blood cells collected with leukapheresis no. 3 will be frozen and stored for possible future use.

Six final vaccines will be given at monthly intervals to further amplify the anti-myeloma white blood cells.

ELIGIBILITY:
Inclusion Criteria:

* MM patients who have active, symptomatic myeloma, and meet the criteria below thus establishing the presence of high-risk myeloma
* MM Salmon-Durie Stage: IA&B (with abnormal cytogenetics*), IIA, IIB, IIIA, and IIIB, and meet the criteria below thus establishing the presence of high-risk myeloma
* MM must meet one of the following criteria: a) Patients who have MAGE-A3 positive MM and who have the tissue type HLA-A*0101, or -* B35, are allocated to receive the MAGE-A3168-176 peptide vaccine. b) Patients who have NY-ESO-1 positive MM and who have the tissue type HLA-A*0201 are allocated to the NY-ESO-1156-C165V peptide vaccine. c) Patients who have NY-ESO-1 positive and MAGE-A3 negative or positive MM and who have as tissue type HLA-A*0101, or -* B35 and HLA-A*0201, will receive vaccination with the NY-ESO-1156-C165V peptide vaccine. d) Patients who have NY-ESO-1 negative and MAGE-A3 positive MM and who have as tissue type HLA-A*0101, or -* B35 and HLA-A*0201, will receive vaccination with the MAGE-A3 peptide vaccine.
* Karnofsky performance score ≥=70, unless bone pain caused by MM results in a Karnofsky score of > or =50.
* Age 18-70 years old
* Hb > or =8.0gm/dl, ANC > or =1,000/microliters, platelet count > or = 100,000/microliters.
* Patients must have signed an IRB-approved consent form and been informed about the investigational nature of the study
* Negative serology for HIV, Hepatitis C and negative for Hepatitis B surface antigen.
* CD4+ count >400/microliters
* Life expectancy > 6 months
* Negative pregnancy test and females agree to two forms of contraception or abstinence.
* Provisional insurance approval for single or double auto-transplant(s)

Exclusion Criteria:

* MGUS, indolent and smoldering myeloma
* Chemotherapy or other immunosuppressive treatment e.g. gluco-corticosteroids, cyclophosphamide, methotrexate within the 4 weeks prior to enrollment
* Patients who have malignancies other than carcinoma-in-situ of the cervix or non-melanomatous skin cancer
* Fever or active infection
* Liver function: total bilirubin > 2.5xULN or AST/ALT >2.5xULN
* Renal function: patients on dialysis, or serum creatinine >2.0mg/dl
* Simultaneous treatment with a second investigational drug or biologic agent for MM
* Other intercurrent serious illness, e.g. cardiac, pulmonary, hepatic disease, uncontrolled diabetes, etc
* Cardiac: Patients with recent (< or =6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrythmias are ineligible. Ejection fraction by ECHO or must be > or = 50% and must be performed within 60 days prior to registration, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the LVEF must be repeated
* Pulmonary: Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease resulting in unacceptable lung function: patients must have adequate pulmonary function studies > or = 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > or = 50% of predicted. Patients unable to complete pulmonary function tests due to myeloma related pain or fracture must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70
* Patients must be able to receive full doses of DT PACE, in the opinion of the treating investigator, with the exception of: A) Patients that have received prior adriamycin > 450 mg/m2 and LVEF < 55%. Adriamycin will be omitted in these patients. B) Patients with a creatinine clearance 30 - 50 ml/minute, who will receive 50% of the cisplatin dose

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, M.D., Ph.D., Principal Investigator — Myeloma Institute for Research & Therapy
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients of the Myeloma Institute who have "high-risk" multiple myeloma because of abnormalities in their cytogenetics, could participate in this study at UAMS only. Final IRB approval was 6/14/04. The 1st participant was enrolled 4/4/05.
Pre-assignment Details: Pre-study: hemogram, blood chemistry, Helper/Suppressor Panel, Immunoknow count, serum protein electrophoresis and immunofixation , serum freelites, 24-hr urine (protein and immunofixation), quantitation of immunoglobulins, B2M, IL6, bone marrow aspiration and biopsy, MRI, bone marrow collection for gene-array.
Groups:
- MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY: Treatment will consist of receiving peptide (small pieces of proteins)vaccinations as a shot just under the skin (subcutaneous). We have chosen to vaccinate with peptides derived from cancer proteins found in myeloma and other cancers. Purpose: to generate anti-myeloma T-cells which will kill only myeloma cells.
  MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY : 3 injections with 300µg/injection (in 1.5mls) of peptide will be given subcutaneously together with the adjuvant GM-CSF at 500µg (same site in 0.5 mls) at two-week intervals.
  MAGE-A3 : vaccinations at 2-week intervals (days 22,36,50) with the MAGE-A3 or NY-ESO-1 peptide and GM-CSF adjuvant. The peptides will be given s.c. in a dose of 300μg; GM-CSF (250μg) will be administered to promote attraction, maturation and longevity of DCs. #2 will be thawed and re-infused after transplant on day 81 and any anti-myeloma T-cells in this leukapheresis product will be boosted immediately by re-vaccinating.
Period: Overall Study
Arm/Group | MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY
Started | 4
Completed | 2
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY: Treatment will consist of receiving peptide (small pieces of proteins) vaccinations as a shot just under the skin (subcutaneous). Purpose is to generate anti-myeloma T-cells with will kill only myeloma cells. Three injections of peptide will be given subcutaneously together with the adjuvant GM-CSF at 2-week intervals.
Arm/Group | MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing a Response to the Peptide Vaccines.
Description: The peptides are fragments from two proteins MAGE-A3 and NY-ESO-1. There will be a series of 12 peptide vaccinations given as a subcutaneous (beneath the skin) injection (vaccines) at 2 week intervals resulting in an immune response to myeloma. The tumor peptides used in the vaccines are unique to myeloma, and it is not expected that there will be an immune response to normal organs. Myeloma cells must express MAGE-A3 or NY-ESO-1, be severe enough to require chemotherapy and stem cell transplantation and have appropriate HLA tissue type.
Time Frame: 2 week intervals
Population: only 2 were complete per protocol. 2 were withdrawn by physician due to relapse.
Measure: Number; unit: participants
Arm/Group | MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY
Number analyzed (Participants) | 4
participants | 2

ADVERSE EVENTS:
Arm/Group | MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAGE-A3 AND NY-ESO-1 IMMUNOTHERAPY (N=4)
DVT (Vascular disorders) | 3 (3)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1)
Staphyloccocal infections (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No